CLINICAL TRIAL: NCT00001036
Title: Safety and Efficacy of Polyethylene Glycolated IL-2 (PEG IL-2) Plus Zidovudine and Thymosin Alpha 1 in HIV-Positive, Asymptomatic and Symptomatic Individuals
Brief Title: The Safety and Effectiveness of a Type of Interleukin-2 Plus Zidovudine Plus Thymosin in HIV-Positive Patients With and Without Symptoms of Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Purpose: Treatment
Other Study IDs: ACTG 236
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-07-30 (Estimated); Status verified 1996-10

CONDITIONS: HIV Infections
Keywords: T-Lymphocytes; Polyethylene Glycols; Interleukin-2; Drug Therapy, Combination; Adjuvants, Immunologic; Acquired Immunodeficiency Syndrome; Zidovudine; thymosin alpha(1)
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Thymalfasin; Interleukin-2; Zidovudine

INTERVENTIONS:
Drug: Thymalfasin
Drug: Interleukin-2, Polyethylene Glycolated
Drug: Zidovudine

SUMMARY:
To determine the safety of thymosin alpha 1 given twice weekly in a regimen of daily oral zidovudine (AZT) and biweekly polyethylene glycolated interleukin-2 (PEG IL-2). To determine the effect of thymosin alpha 1 and PEG IL-2 in combination with AZT on immunologic and pharmacokinetic markers.

AIDS is characterized by diminished T helper cell number and function. Thymosin alpha 1 appears to both increase IL-2 receptors on lymphocytes in vitro and enhance lymphocyte maturation in vivo; thus, the drug may further enhance the CD4 T cell levels in patients receiving AZT and PEG IL-2.

DETAILED DESCRIPTION:
AIDS is characterized by diminished T helper cell number and function. Thymosin alpha 1 appears to both increase IL-2 receptors on lymphocytes in vitro and enhance lymphocyte maturation in vivo; thus, the drug may further enhance the CD4 T cell levels in patients receiving AZT and PEG IL-2.

Patients are stabilized on oral AZT daily for 8 weeks and then begin receiving bolus infusions of PEG IL-2 every other week for at least four doses. Thymosin alpha 1 (given SC) is then added to this regimen twice weekly for 4 weeks. If no significant toxicity occurs, thymosin alpha 1 is increased to and administered along with scheduled doses of PEG IL-2 for an additional 8 weeks.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Prophylactic pentamidine for Pneumocystis carinii.

Patients must have:

* HIV seropositivity.
* CD4 count > 50 and < 200 cells/mm3.
* No active opportunistic infections.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Concurrent neoplasms other than basal cell carcinoma of the skin, in situ carcinoma of the cervix, or Kaposi's sarcoma.
* Significant cardiac disease or CNS lesions or other neurologic abnormalities.
* Score of > 0.5 on ACTG AIDS Dementia Complex staging.
* Major organ allograft.
* Intolerance to AZT at 500 mg/day.

Concurrent Medication:

Excluded:

* Antihypertensive medication other than diuretics.
* Chemotherapy, hormonal therapy, or other immunotherapy.
* Other investigational drugs, agents, or devices.
* Beta-blockers.
* Non-topical steroids.

Concurrent Treatment:

Excluded:

* Radiation therapy.

Prior Medication:

Excluded:

* Known anti-HIV medication (other than AZT) or known immunomodulators (e.g., systemic steroids, interferons, interleukins) or other chemotherapy within 30 days prior to study entry.

Prior Treatment:

Excluded:

* Transfusion within 4 weeks prior to study entry.
* Radiation within 30 days prior to study entry.

Active substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12

CONTACTS AND LOCATIONS:
Overall Officials: TC Merigan, Study Chair
Locations (1):
- Stanford Univ Med Ctr, Stanford, California, United States

REFERENCES:
- [Background] Ramachandran R, Katzenstein DA, Winters MA, Kundu SK, Merigan TC. Polyethylene glycol-modified interleukin-2 and thymosin alpha 1 in human immunodeficiency virus type 1 infection. J Infect Dis. 1996 Apr;173(4):1005-8. doi: 10.1093/infdis/173.4.1005. PMID 8603940